CLINICAL TRIAL: NCT00571727
Title: A Study of Long-Term Human Recombinant Insulin-Like Growth Factor-1 (rhIGF-1) in Children With Short Stature Due to Growth Hormone Insensitivity Syndrome (GHIS)
Brief Title: Long-Term Treatment With rhIGF-1 in GHIS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Collaborators: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Study 1419
Record Dates: First submitted 2007-12-10; First posted 2007-12-12 (Estimated); Results first posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Growth Hormone Insensitivity Syndrome
Keywords: growth; insulin like growth factor; Laron syndrome
MeSH Terms: conditions — Laron Syndrome | interventions — mecasermin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

ARMS (1):
- mecasermin, injections BID of rhIGF-1 (Experimental)
  Interventions: Drug: mecasermin

INTERVENTIONS:
Drug: mecasermin — injections BID of rhIGF-1, mecasermin
  Other Names: Increlex

SUMMARY:
The objective of this study was to evaluate the long-term safety and effectiveness of mecasermin (the study drug) in children with growth failure due to severe Primary insulin-like growth factor-1 deficiency (Primary IGFD).

ELIGIBILITY:
Inclusion Criteria:

* Height <-2SD for age and gender
* IGF-1 <-2SD for age and gender
* Evidence of GH resistance

Exclusion Criteria:

* closed epiphyses
* prior active malignancy
* major organ disfunction
* treatment with medications that would diminish growth
* clinically significant cardiac abnormalities

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 92 (Actual)
Dates: Start 1991-05-20 (Actual); Primary Completion 2011-12-15 (Actual); Study Completion 2011-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (1):
- Ipsen, Brisbane, California, United States

REFERENCES:
- [Result] Chernausek SD, Backeljauw PF, Frane J, Kuntze J, Underwood LE; GH Insensitivity Syndrome Collaborative Group. Long-term treatment with recombinant insulin-like growth factor (IGF)-I in children with severe IGF-I deficiency due to growth hormone insensitivity. J Clin Endocrinol Metab. 2007 Mar;92(3):902-10. doi: 10.1210/jc.2006-1610. Epub 2006 Dec 27. PMID 17192294

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 3, open-label study was conducted in children with short stature due to severe primary insulin like growth factor-1 deficiency at 2 investigative sites in the US in conjunction with sites in 23 other countries (Argentina, Australia, Austria, Bahamas, Brazil, Canada, Egypt, France, Germany, Iran, Israel, Italy, Kuwait, Pakistan, Poland, Russia, Saudi Arabia, Spain, Sweden, Syria, Taiwan, Ukraine, and Yemen).
Pre-assignment Details: Participants who had been treated with mecasermin in previous Genentech-sponsored studies (F0206s, F0375g, F0632g, F0671g), as well as new participants naïve to mecasermin treatment, were enrolled in this study.
Groups:
- Mecasermin: Participants who were entered from previous studies continued to receive mecasermin 80 to 120 microgram per kilograms (mcg/kg) subcutaneously (SC) twice daily and naïve-to-treatment participants were administered mecasermin 60 to 80 mcg/kg SC twice daily for 1 to 2 weeks, and then increased to 120 mcg/kg as tolerated.
Period: Overall Study
Arm/Group | Mecasermin
Started | 92
Completed | 26
Not Completed | 66
Not completed — Did not enter in this study | 1
Not completed — Non-compliance | 4
Not completed — Lost to Follow-up | 30
Not completed — Poor growth | 1
Not completed — Parent/patient decision | 2
Not completed — Participant transferred to commercial drug | 14
Not completed — Unable to provide study drug | 6
Not completed — On-treatment at end of study | 8

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of mecasermin treatment.
Groups:
- Mecasermin: Participants who were entered from previous studies continued to receive mecasermin 80 to 120 mcg/kg SC twice daily and naïve-to-treatment participants were administered mecasermin 60 to 80 mcg/kg SC twice daily for 1 to 2 weeks, and then increased to 120 mcg/kg as tolerated.
Arm/Group | Mecasermin
Number analyzed (Participants) | 92
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.6 (4.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 53
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 77
  African American | 3
  Hispanic | 6
  Asian | 4
  Other | 2

OUTCOME MEASURES:

1. Primary Outcome: Annualized Height Velocity Up to 12 Years
Description: Height velocity is the difference between 2 height measurements, divided by years elapsed between measurements.
Time Frame: Baseline (Pre-dose) and up to 12 years
Population: The intention-to-treat population consisted of all 92 participants. Only data from the participants naïve to exogenous recombinant human insulin-like growth factor-1 (rhIGF-1) and whose pre-treatment height velocity were available were reported.
Measure: Mean (Standard Deviation); unit: centimeter per year (cm/y)
Arm/Group | Mecasermin
Number analyzed (Participants) | 75
centimeter per year (cm/y)
  Baseline (Pre-dose) | 2.6 (1.7)
  >= 1 year | 8.0 (2.3)
  >= 2 years: number analyzed (Participants) | 63
  >= 2 years | 5.9 (1.7)
  >= 3 years: number analyzed (Participants) | 62
  >= 3 years | 5.5 (1.8)
  >= 4 years: number analyzed (Participants) | 60
  >= 4 years | 5.2 (1.5)
  >= 5 years: number analyzed (Participants) | 53
  >= 5 years | 4.9 (1.5)
  >= 6 years: number analyzed (Participants) | 39
  >= 6 years | 4.8 (1.4)
  >= 7 years: number analyzed (Participants) | 25
  >= 7 years | 4.3 (1.5)
  >= 8 years: number analyzed (Participants) | 19
  >= 8 years | 4.4 (1.5)
  >= 9 years: number analyzed (Participants) | 14
  >= 9 years | 4.4 (1.7)
  >= 10 years: number analyzed (Participants) | 13
  >= 10 years | 4.5 (2.0)
  >= 11 years: number analyzed (Participants) | 12
  >= 11 years | 4.1 (2.0)
  >= 12 years: number analyzed (Participants) | 10
  >= 12 years | 3.9 (2.0)

2. Primary Outcome: Number of Naive Participants With Height Velocity <5 cm/y at the End of 1 Year of Study Treatment
Description: Height measurements were performed using wall-mounted stadiometers for analysis of growth data.
Time Frame: Baseline (Pre-dose) and 1 year
Population: The intention-to-treat population consisted of all 92 participants. Only data from the participants naïve to exogenous rhIGF-1 were reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Mecasermin
Number analyzed (Participants) | 81
Participants | 7

3. Secondary Outcome: Height Velocity Standard Deviation Score Up to 12 Years
Description: Center for disease control growth charts from the US were used as reference for age and gender-dependent mean and standard deviation. Height velocity-standard deviation score was calculated as height velocity minus reference mean height velocity divided by standard deviation of the reference mean height velocity. Greater height velocity standard deviation score indicates better outcome.
Time Frame: Baseline (Pre-dose) and up to 12 years
Population: The intention-to-treat population consisted of all 92 participants. Only data from the participants naïve to exogenous rhIGF-1 and whose pre-treatment height velocity were available were reported.
Measure: Mean (Standard Deviation); unit: Standard deviation score
Arm/Group | Mecasermin
Number analyzed (Participants) | 75
Standard deviation score
  Baseline (Pre-dose) | -3.4 (1.6)
  >= 1 year | 1.7 (2.8)
  >= 2 years: number analyzed (Participants) | 62
  >= 2 years | -0.0 (1.7)
  >= 3 years: number analyzed (Participants) | 61
  >= 3 years | -0.1 (1.9)
  >= 4 years: number analyzed (Participants) | 58
  >= 4 years | -0.2 (1.9)
  >= 5 years: number analyzed (Participants) | 50
  >= 5 years | -0.3 (1.7)
  >= 6 years: number analyzed (Participants) | 37
  >= 6 years | -0.2 (1.6)
  >= 7 years: number analyzed (Participants) | 22
  >= 7 years | -0.5 (1.7)
  >= 8 years: number analyzed (Participants) | 15
  >= 8 years | -0.2 (1.6)
  >= 9 years: number analyzed (Participants) | 12
  >= 9 years | -0.4 (0.8)
  >= 10 years: number analyzed (Participants) | 11
  >= 10 years | 0.1 (1.6)
  >= 11 years: number analyzed (Participants) | 11
  >= 11 years | 0.5 (2.6)
  >= 12 years: number analyzed (Participants) | 8
  >= 12 years | -0.1 (1.5)

4. Secondary Outcome: Height Standard Deviation Score Up to 12 Years
Description: Center for disease control growth charts from the US were used as reference for age and gender-dependent mean and standard deviation. Height standard deviation score was calculated as height minus reference mean height divided by standard deviation of the reference mean height. A higher height standard deviation score indicates a better outcome.
Time Frame: Baseline (Pre-dose) and up to 12 years
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Standard deviation score
Arm/Group | Mecasermin
Number analyzed (Participants) | 81
Standard deviation score
  Baseline (Pre-dose) | -6.9 (1.8)
  >= 1 year | -6.1 (1.8)
  >= 2 years: number analyzed (Participants) | 67
  >= 2 years | -5.6 (1.7)
  >= 3 years: number analyzed (Participants) | 66
  >= 3 years | -5.3 (1.7)
  >= 4 years: number analyzed (Participants) | 64
  >= 4 years | -5.1 (1.7)
  >= 5 years: number analyzed (Participants) | 57
  >= 5 years | -5.0 (1.7)
  >= 6 years: number analyzed (Participants) | 41
  >= 6 years | -4.9 (1.6)
  >= 7 years: number analyzed (Participants) | 26
  >= 7 years | -4.9 (1.7)
  >= 8 years: number analyzed (Participants) | 19
  >= 8 years | -5.1 (1.7)
  >= 9 years: number analyzed (Participants) | 14
  >= 9 years | -5.0 (1.6)
  >= 10 years: number analyzed (Participants) | 13
  >= 10 years | -5.0 (1.7)
  >= 11 years: number analyzed (Participants) | 12
  >= 11 years | -4.7 (1.2)
  >= 12 years: number analyzed (Participants) | 10
  >= 12 years | -4.4 (1.3)

5. Secondary Outcome: Approximate Increase in Height Over Expected for Naïve Participants With Near-Adult Height
Description: Height measurements were performed using wall-mounted stadiometers for analysis of growth data.
Time Frame: Baseline (Pre-dose) and up to 19 years
Population: The intention-to-treat population consisted of all 92 participants. Only data from the participants naïve to exogenous rhIGF-1 and who attained near adult height were reported.
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Mecasermin
Number analyzed (Participants) | 21
cm | 13.3 (8.4)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events were collected from first date of mecasermin intake until last dose, approximately 19 years
Description: The safety population consisted of all participants who had received at least 1 dose of mecasermin treatment. Adverse events were not collected per dose level as pre-specified.
Arm/Group | Mecasermin
All-Cause Mortality (participants affected / at risk) | 0/92
Serious Adverse Events (participants affected / at risk) | 18/92
Other Adverse Events (participants affected / at risk) | 73/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mecasermin (N=92)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Infectious pleural effusion (Infections and infestations) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1)
Appendicitis (Infections and infestations) | 2 (2)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Benign intracranial hypertension (Nervous system disorders) | 1 (1)
Epiphysiolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Dilatation ventricular (Cardiac disorders) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Febrile convulsion (Nervous system disorders) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Hypoglycaemic seizure (Metabolism and nutrition disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mecasermin (N=92)
Hypoglycaemia (Metabolism and nutrition disorders) | 41 (175)
Hypoglycaemic seizure (Metabolism and nutrition disorders) | 5 (13)
Injection site hypertrophy (General disorders) | 32 (211)
Pyrexia (General disorders) | 19 (77)
Fatigue (General disorders) | 9 (16)
Injection site haematoma (General disorders) | 9 (22)
Hypertrophy (General disorders) | 8 (52)
Asthenia (General disorders) | 5 (7)
Chest pain (General disorders) | 5 (10)
Upper respiratory tract infection (Infections and infestations) | 23 (73)
Otitis media (Infections and infestations) | 19 (76)
Nasopharyngitis (Infections and infestations) | 14 (36)
Influenza (Infections and infestations) | 12 (17)
Bronchitis (Infections and infestations) | 7 (8)
Ear infection (Infections and infestations) | 7 (19)
Gastroenteritis (Infections and infestations) | 7 (9)
Pharyngitis (Infections and infestations) | 7 (16)
Respiratory tract infection (Infections and infestations) | 6 (7)
Tonsillitis (Infections and infestations) | 6 (8)
Varicella (Infections and infestations) | 5 (5)
Snoring (Respiratory, thoracic and mediastinal disorders) | 20 (111)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 19 (102)
Cough (Respiratory, thoracic and mediastinal disorders) | 16 (48)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 7 (12)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9 (37)
Vomiting (Gastrointestinal disorders) | 16 (28)
Dental caries (Gastrointestinal disorders) | 11 (45)
Abdominal pain (Gastrointestinal disorders) | 7 (13)
Constipation (Gastrointestinal disorders) | 6 (10)
Diarrhoea (Gastrointestinal disorders) | 6 (14)
Abdominal pain upper (Gastrointestinal disorders) | 5 (6)
Tooth crowding (Gastrointestinal disorders) | 5 (24)
Toothache (Gastrointestinal disorders) | 5 (11)
Headache (Nervous system disorders) | 25 (109)
Dizziness (Nervous system disorders) | 6 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (24)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 (25)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (18)
Acne (Skin and subcutaneous tissue disorders) | 10 (26)
Dry skin (Skin and subcutaneous tissue disorders) | 10 (31)
Skin hypertrophy (Skin and subcutaneous tissue disorders) | 10 (36)
Rash (Skin and subcutaneous tissue disorders) | 6 (9)
Conductive deafness (Ear and labyrinth disorders) | 11 (70)
Middle ear effusion (Ear and labyrinth disorders) | 10 (21)
Deafness (Ear and labyrinth disorders) | 6 (50)
Ear pain (Ear and labyrinth disorders) | 6 (9)
Ear discomfort (Ear and labyrinth disorders) | 5 (27)
Cardiac murmur (Investigations) | 7 (10)
Thymus enlargement (Blood and lymphatic system disorders) | 9 (24)
Lymphadenopathy (Blood and lymphatic system disorders) | 5 (9)
Papilloedema (Eye disorders) | 5 (7)
Tachycardia (Cardiac disorders) | 6 (6)
Gynaecomastia (Reproductive system and breast disorders) | 6 (18)
Ear tube insertion (Surgical and medical procedures) | 7 (11)
Dental operation (Surgical and medical procedures) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other